CLINICAL TRIAL: NCT01439971
Title: An Ascending Single Dose Study To Evaluate The Safety, Tolerability And Pharmacokinetics/Pharmacodynamics Of Pf-05280602, A Recombinant Factor Viia Variant (813d), In Adult Hemophilia A And B Subjects With Or Without Inhibitors
Brief Title: Phase 1 Safety, Pharmacokinetics And Pharmacodynamics Study Of Recombinant Factor VIIa Variant (813d) In Adult Subjects With Hemophilia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catalyst Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: B3051001; 2011-002170-23 (EudraCT Number)
Record Dates: First submitted 2011-08-26; First posted 2011-09-23 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Hemophilia A
Keywords: Phase 1; Safety; Pharmacokinetic; Pharmacodynamic
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Intervention Model Description: The was an ascending dose trial with one open label treatment, intervention model was sequential dose escalation.
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental)
  Interventions: Biological: PF-05280602
- 2 (Experimental)
  Interventions: Biological: PF-05280602
- 3 (Experimental)
  Interventions: Biological: PF-05280602
- 4 (Experimental)
  Interventions: Biological: PF-05280602
- 5 (Experimental)
  Interventions: Biological: PF-05280602

INTERVENTIONS:
Biological: PF-05280602 — 0.5 micrograms per kilogram of PF-05280602, IV infusion, single dose
  Arms: 1
Biological: PF-05280602 — 4.5 micrograms per kilogram of PF-05280602, IV infusion, single dose
  Arms: 2
Biological: PF-05280602 — 9.0 micrograms per kilogram of PF-05280602, IV infusion, single dose
  Arms: 3
Biological: PF-05280602 — 18.0 micrograms per kilogram of PF-05280602, IV infusion, single dose
  Arms: 4
Biological: PF-05280602 — 30.0 micrograms per kilogram of PF-05280602, IV infusion, single dose
  Arms: 5

SUMMARY:
This study hypothesizes that the study drug, PF-05280602 (at the selected doses) will be safe to administer to subjects with severe Hemophilia A or B with or without inhibitors and will demonstrate evidence of hemostatic activity. This is supported by the preclinical findings in hemophilic animal models.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects 18 to <65 years old with severe hemophilia A or B with or without inhibitors to FVIII or FIX.
* Subjects is willing and able to comply with the mandatory washout periods prior to screening and prior to dosing and through 48 hours post dosing. At screening this includes a washout of FIX for 96 hours and FVIII for 72 houts. At dosing this includes a washout of FIX for 96 hours and FVIII and other hemostatic agents for 72 hours through 48 hours post dosing.
* Subjects must agree and commit to using a a highly effective method of birth control from the time of screening through four weeks after study drug administration.

Exclusion Criteria:

* Presence of a bleeding disorder in addition to hemophilia A or B.
* Regular, concomitant therapy with immunomodulating drugs (eg, intravenous immunoglobulin, and routine systemic corticosteroids).
* History of coronary artery disease, thrombolic disease or diagnosis of prothrombic disorder.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- United States (9):
  - University of California San Diego Medical Center, San Diego, California
  - New Haven Clinical Research Unit, New Haven, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - OHSU Investigational Pharmacy, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - CTRC, Philadelphia, Pennsylvania
  - Penn Comprehensive Hemophilia Program - Center for Blood Disorders, Philadelphia, Pennsylvania
- Pfizer Clinical Research Unit, Brussels, Belgium
- Semmelweis Egyetem Altalanos Orvostudomanyi Kar/ I.sz. Belgyogyaszati Klinika, Budapest, Hungary
- Italy (6):
  - Dipartimento di Medicina Clinica 1-Centro Regionale per le Malattie del Sangue, Castelfranco Veneto (TV), Italy
  - Servizio Farmacia- Ospedale Castelfranco Veneto, Castelfranco Veneto - Treviso, Italy
  - Servizio Farmacia Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy
  - Farmacia Ospedaliera Ospedale San Bortolo, Vicenza, Italy
  - Centro Emofilia e Trombosi "Angelo Bianchi Bonomi" U.O.S. Dipartimentale per la Diagnosi e la Terapi, Milan
  - Centro Malattie Emorragiche e Trombotiche - Ematologia, Vicenza
- Christchurch Clinical Studies Trust, Christchurch, New Zealand, New Zealand
- Phoenix Pharma (Pty) Ltd, Port Elizabeth, Eastern Cape, South Africa
- Ege University Tip Fakultesi, Izmir, Turkey, Turkey (Türkiye)
- United Kingdom (3):
  - Royal Free Hampstead NHS Trust, Royal Free Hospital, London
  - Haematology Department, London
  - Central Manchester Universtiy Hospitals NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3051001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label study to characterize the single dose pharmacokinetics (PK), pharmacodynamics, safety, and tolerability of 5 intravenous dose levels of PF-05280602 (0.5, 4.5, 9.0, 18.0 and 30.0 micrograms/kilogram [mcg/kg]).
Groups:
- PF-05280602 0.5 mcg/kg: PF-05280602 0.5 mcg/kg, the original lowest dosing arm, was administered as a single dose of bolus intravenous infusion on Day 1. The protocol was amended after a single participant was enrolled and the starting dose was changed to 4.5 mcg/kg.
- PF-05280602 4.5 mcg/kg: PF-05280602 4.5 mcg/kg was administered as a single dose of bolus intravenous infusion on Day 1.
- PF-05280602 9.0 mcg/kg: PF-05280602 9.0 mcg/kg was administered as a single dose of bolus intravenous infusion on Day 1.
- PF-05280602 18.0 mcg/kg: PF-05280602 18.0 mcg/kg was administered as a single dose of bolus intravenous infusion on Day 1.
- PF-05280602 30.0 mcg/kg: PF-05280602 30.0 mcg/kg was administered as a single dose of bolus intravenous infusion on Day 1.
Period: Overall Study
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Started | 1 | 7 | 8 | 6 | 7
Received Treatment | 1 | 6 | 6 | 6 | 6
Completed | 1 | 6 | 6 | 6 | 6
Not Completed | 0 | 1 | 2 | 0 | 1
Not completed — Required number in cohort dosed | 0 | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all enrolled participants who received the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg | Total
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (NA) — Single participant in cohort | 32.7 (13.4) | 38.5 (12.1) | 32.8 (12.3) | 41.0 (15.7) | 37.2 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 0 | 0 | 0 | 0 | 0 | 0
  MALE | 1 | 6 | 6 | 6 | 6 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Supine blood pressure (BP) was measured with the participant's arm supported at the level of the heart, and recorded to the nearest millimeters of mercury (mmHg) after 5 minutes of rest. The same arm (preferably the dominant arm) was to be used throughout the study.
Time Frame: Baseline, Day 2, Day 3, and Day 15
Population: The safety population included all enrolled participants who received the study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
mmHg
  SBP: Baseline | 122.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 130.2 (7.14) | 120.2 (25.41) | 124.2 (7.68) | 125.5 (8.53)
  SBP: Change at Day 2 | 0.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | -8.7 (8.24) | -0.2 (14.41) | -3.0 (6.51) | -1.5 (5.58)
  SBP: Change at Day 3 | 5.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | -7.0 (6.99) | 2.2 (19.30) | -5.5 (7.66) | 0.0 (8.58)
  SBP: Change at Day 15 | -10.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | -5.5 (12.18) | 4.7 (18.00) | -4.5 (14.92) | 1.8 (11.84)
  DBP: Baseline | 78.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 73.7 (6.35) | 70.5 (10.97) | 75.8 (4.67) | 77.0 (6.87)
  DBP: Change at Day 2 | 2.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | -2.8 (6.43) | 2.7 (6.28) | -0.8 (5.12) | -3.3 (5.50)
  DBP: Change at Day 3 | -3.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | -6.5 (6.57) | 3.3 (6.56) | -2.2 (8.11) | 4.3 (10.41)
  DBP: Change at Day 15 | -9.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | -3.5 (11.41) | 6.0 (13.11) | -4.3 (11.15) | -4.5 (5.65)

2. Primary Outcome: Change From Baseline in Body Weight
Time Frame: Baseline, Day 2, Day 3, and Day 15
Population: The safety population included all enrolled participants who received the study drug.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
kilograms (kg)
  Baseline | 72.7 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 75.0 (12.65) | 78.7 (10.73) | 78.0 (11.31) | 73.4 (6.88)
  Change at Day 2 | -0.9 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | -1.0 (0.98) | -0.6 (0.72) | -0.8 (1.31) | -0.4 (0.83)
  Change at Day 3 | -0.8 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | -0.6 (0.85) | -0.5 (0.60) | -0.8 (1.39) | -0.3 (0.56)
  Change at Day 15 | -0.5 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 0.4 (1.09) | 0.6 (1.55) | 0.6 (1.26) | 0.2 (0.59)

3. Primary Outcome: Change From Baseline in Body Temperature
Description: Body temperature was measured by mouth (oral) or ear (tympanic). A temperature greater than 38.5 degree Celsius was considered a fever.
Time Frame: Baseline, Day 2, Day 3, and Day 15
Population: The safety population included all enrolled participants who received the study drug.
Measure: Mean (Standard Deviation); unit: degree Celcius
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
degree Celcius
  Baseline | 36.1 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 36.5 (0.29) | 36.5 (0.34) | 36.6 (0.30) | 36.4 (0.43)
  Change at Day 2 | 0.4 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | -0.4 (0.62) | -0.1 (0.30) | 0.1 (0.34) | 0.2 (0.29)
  Change at Day 3 | 0.3 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | -0.2 (0.60) | 0.1 (0.15) | -0.0 (0.41) | 0.2 (0.13)
  Change at Day 15 | 0.3 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 0.1 (0.39) | 0.1 (0.36) | 0.1 (0.24) | 0.2 (0.60)

4. Primary Outcome: Change From Baseline in Respiration Rate
Description: Respiration rate measured as respirations per minute (resp/min).
Time Frame: Baseline, Day 2, Day 3, and Day 15
Population: The safety population included all enrolled participants who received the study drug.
Measure: Mean (Standard Deviation); unit: resp/min
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
resp/min
  Baseline | 12.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 15.0 (2.76) | 15.2 (2.04) | 15.7 (1.97) | 16.0 (2.83)
  Change at Day 2 | 0.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 0.5 (1.76) | 0.3 (3.50) | 2.2 (2.56) | 0.5 (1.22)
  Change at Day 3 | 0.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 0.2 (3.37) | 0.3 (3.50) | 1.7 (1.63) | 0.2 (2.23)
  Change at Day 15 | 2.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 0.7 (4.32) | -0.2 (2.14) | 1.2 (3.49) | -0.3 (1.97)

5. Primary Outcome: Change From Baseline in Supine Pulse Rate
Description: Change from baseline is the vital sign value at Day 2, Day 3, and Day 15 minus vital sign value at baseline.
Time Frame: Baseline, Day 2, Day 3, and Day 15
Population: The safety population included all enrolled participants who received the study drug.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
beats per minute (bpm)
  Baseline | 62.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 64.8 (6.21) | 69.3 (10.65) | 60.7 (10.69) | 66.5 (8.22)
  Change at Day 2 | 1.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | -1.3 (3.56) | 3.7 (6.89) | 8.8 (7.88) | 2.0 (5.69)
  Change at Day 3 | 0.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 1.3 (6.80) | 2.5 (7.89) | 10.7 (5.65) | 3.3 (3.56)
  Change at Day 15 | 2.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 8.3 (12.68) | 4.5 (12.68) | 10.2 (12.22) | 3.0 (5.33)

6. Primary Outcome: Number of Participants With Changes Since Previous Physical Examination
Description: Physical examinations were conducted by a physician, trained physician's assistant, or nurse practitioner. A complete physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, genitourinary, gastrointestinal, musculoskeletal, and neurological systems. The limited or abbreviated physical examination focused on general appearance, the respiratory and cardiovascular systems, as well as towards participant reported symptoms.
Time Frame: Baseline (Day 0), Day 1, Day 2, Day 3, Day 15
Population: The safety population included all enrolled participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
participants
  Baseline | 0 | 0 | 0 | 0 | 0
  Day 1 | 0 | 0 | 0 | 0 | 0
  Day 2 | NA — No participants were analyzed at Day 2 in this arm. | 0 | 1 | 0 | 0
  Day 3 | 0 | 0 | 1 | 1 | 0
  Day 15 | 0 | 1 | 0 | 1 | 0

7. Primary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Findings
Description: ECG findings of potential clinical concern were: PR interval greater than or equal to (>=)300 milliseconds (msec), >=25% increase from baseline for baseline values >200 msec, >=50% increase from baseline for baseline values less than or equal to (<=)200 msec; QRS complex >=140 msec or >=50% increase from baseline; QTcF interval (Fridericia's correction) >=450 msec or >=30 msec increase from baseline.
Time Frame: Baseline through Day 15
Population: The safety population included all enrolled participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
participants
  PR Interval >=300 msec | 0 (NA) | 0 (7.14) | 0 (25.41) | 0 (7.68) | 0 (8.53)
  QRS Complex >=140 msec | 0 | 0 | 0 | 0 | 0
  QTcF Interval >=450 msec | 0 | 0 | 0 | 0 | 0
  PR Interval >=25/50% Increase From Baseline | 0 | 0 | 0 | 0 | 0
  QRS Complex >=50% Increase From Baseline | 0 | 0 | 0 | 0 | 0
  QTcF Interval 30-<60 msec Increase From Baseline | 0 | 1 | 0 | 0 | 0
  QTcF Interval >=60 msec Increase From Baseline | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs), and Withdrawals Due to AEs (Except Hemophilia AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Day 15 that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline through Day 60
Population: The safety population included all enrolled participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
participants
  AEs | 1 | 4 | 4 | 3 | 2
  SAEs | 0 | 0 | 0 | 0 | 0
  Withdrawals Due to AEs | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Treatment-Emergent Hemophilia AEs and Withdrawals Due to Hemophilia AEs
Description: Hemophilia AEs included spontaneous (no known contributing factor) and traumatic (known or presumed contributing factor/reason) bleeding episodes.
Time Frame: Baseline through Day 60
Population: The safety population included all enrolled participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
participants
  Hemophilia AEs | 1 | 1 | 1 | 1 | 2
  Hemophilia SAEs | 0 | 0 | 0 | 0 | 0
  Withdrawals Due to Hemophilia AEs | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Treatment-Emergent AEs and SAEs by Severity (Except Hemophilia AEs)
Description: AE severity were graded as mild, moderate, or severe. Mild severity AEs do not interfere with the participant's usual function. Moderate AEs interfere to some extent with the participant's usual function. Severe AEs interfere significantly with the participant's usual function.
Time Frame: Baseline through Day 60
Population: The safety population included all enrolled participants who received the study drug.
Measure: Number; unit: adverse events
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
adverse events
  Mild AEs | 2 | 6 | 5 | 7 | 1
  Moderate AEs | 1 | 1 | 5 | 2 | 1
  Severe AEs | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Treatment-Emergent Hemophilia AEs by Severity
Description: Mild severity AEs do not interfere with the participant's usual function. Moderate AEs interfere to some extent with the participant's usual function. Severe AEs interfere significantly with the participant's usual function.
Time Frame: Baseline through Day 60
Population: The safety population included all enrolled participants who received the study drug.
Measure: Number; unit: adverse events
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
adverse events
  Mild Hemophilia AEs | 1 | 0 | 0 | 0 | 0
  Moderate Hemophilia AEs | 1 | 1 | 2 | 1 | 2
  Severe Hemophilia AEs | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Treatment-Emergent Abnormal Troponin-T Levels by Magnitude
Description: Troponin-T is a cardiac marker for the evaluation of possible cardiovascular injury. Troponin-T levels of potential clinical concern are values >1.5 times the upper limit of normal (1.5X ULN) or >=2.5X ULN.
Time Frame: Baseline through Day 15
Population: The safety population included all enrolled participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
participants
  <1X lower limit of normal (LLN) | 0 | 0 | 0 | 0 | 0
  >1X ULN | 0 | 0 | 0 | 0 | 0
  >1.5X ULN | 0 | 0 | 0 | 0 | 0
  >=2.5X ULN | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Treatment-Emergent Abnormal Anti-Thrombin III (ATIII) Levels by Magnitude
Description: ATIII is a protein in the blood that blocks abnormal blood clots from forming. Low levels of ATIII can cause abnormal blood clots. ATIII levels of potential clinical concern are values <1X LLN and >1X ULN.
Time Frame: Baseline through Day 3
Population: The safety population included all enrolled participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
participants
  <1X LLN | 0 | 0 | 0 | 0 | 2
  >1X ULN | 0 | 0 | 0 | 1 | 0

14. Primary Outcome: Number of Participants With Treatment-Emergent Abnormal Tissue Factor Pathway Inhibitor (TFPI) Levels by Magnitude
Description: TFPI is a polypeptide that can regulate blood coagulation. TFPI levels of potential clinical concern are values <1X LLN and >1X ULN.
Time Frame: Baseline through Day 3
Population: The safety population included all enrolled participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
participants
  <1X LLN | 0 | 1 | 2 | 0 | 0
  >1X ULN | 1 | 0 | 0 | 0 | 1

15. Primary Outcome: Number of Participants With Treatment-Emergent Laboratory Test Abnormalities (Normal Baseline)
Description: The following laboratory parameters were analyzed: hematology (hemoglobin, hematocrit, red blood cell [RBC] count, platelets, leukocytes, total neutrophils, eosinophils, basophils, lymphocytes, monocytes); chemistry (total bilirubin, direct bilirubin, indirect bilirubin, aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase, creatinine, blood urea nitrogen [BUN], glucose, uric acid, sodium, potassium, chloride, bicarbonate, calcium, albumin, total protein, creatine kinase); urinalysis (urine white blood cell [WBC], urine RBC); other (troponin T).
Time Frame: Baseline through Day 15
Population: The safety population included all enrolled participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
participants | 0 | 0 | 2 | 1 | 2

16. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities Meeting Stopping Criteria
Description: Clinically significant findings for stopping rules are: hemoglobin <8 grams/deciliter (g/dL) or >20% decrease from normal baseline; WBC >20,000 cells/mm^3 or <1,500 decrease with normal baseline; platelets <100,000/mm^3 or >33% decrease from baseline; total bilirubin >1.5X ULN; AST or ALT >2.5X ULN; alkaline phosphatase >3X ULN; creatinine >1.5X baseline; BUN >31.0 mg/dL; glucose <0.6 or >1.5X reference range; uric acid > ULN; sodium >150 or <130 mEq/L; potassium >5.5 or <3.0 mEq/L; calcium >11.5 or <8.0 mg/dL; albumin <2.0 g/L; total protein <5.0 g/L; positive D-dimer at Day 15; PT prolonged by 3 seconds above baseline; ATIII < LLN and >20% decrease from baseline; troponin-T values above the reference range; fibrinogen <0.75X LLN or >25% decrease from baseline.
Time Frame: Baseline through Day 15
Population: The safety population included all enrolled participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
participants
  Hemoglobin | 0 | 0 | 0 | 0 | 0
  Platelets | 0 | 0 | 0 | 0 | 0
  WBC | 0 | 0 | 0 | 0 | 0
  Prothrombin Time | 0 | 0 | 0 | 0 | 0
  Total Bilirubin | 0 | 0 | 0 | 0 | 0
  Total Protein | 0 | 0 | 0 | 0 | 0
  Albumin | 0 | 0 | 0 | 0 | 0
  AST | 0 | 0 | 0 | 0 | 0
  ALT | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase | 0 | 0 | 0 | 0 | 0
  BUN | 0 | 0 | 0 | 0 | 0
  Creatinine | 0 | 1 | 0 | 0 | 0
  Uric Acid | 0 | 0 | 0 | 0 | 0
  Sodium | 0 | 0 | 0 | 0 | 0
  Potassium | 0 | 0 | 1 | 0 | 0
  Calcium | 0 | 0 | 0 | 0 | 0
  Glucose | 0 | 0 | 1 | 1 | 0
  Fibrinogen | 0 | 0 | 0 | 0 | 1
  Troponin-T | 0 | 0 | 0 | 0 | 0
  Anti-Thrombin III | 0 | 0 | 0 | 0 | 0
  D-Dimer | 0 | 0 | 0 | 0 | 1

17. Primary Outcome: Number of Participants With Positive Immune Response (Anti-Drug Antibodies [ADA], PF-05280602 Inhibitor, Factor VIIa Inhibitor, Factor VII Inhibitor, and Depletion of Factor VII Activity)
Description: Assays for the determination of a positive immune response was performed. An antibody immune response was defined as a confirmed post-treatment positive ELISA result in combination with a negative baseline sample ELISA result. Positive antibody immune responses to PF-05280602 by ELISA was evaluated for cross reactivity to NovoSeven RT and to Factor VII.
Time Frame: Baseline through Day 60
Population: The immunogenicity parameter population included enrolled and treated participants with at least 1 post-treatment anti-PF-05280602 antibody (ADA), PF-05280602 inhibitor, or Factor VII activity level determination.
Measure: Number; unit: participants
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
participants
  ADA | 0 | 0 | 0 | 1 | 0
  PF-05280602 Inhibitor | 0 | 0 | 0 | 0 | 0
  Factor VIIa Inhibitor | 0 | 0 | 0 | 0 | 0
  Factor VII Inhibitor | 0 | 0 | 0 | 0 | 0
  Depletion of Factor VII Activity | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Day 1 (pre-dose and 5 min, 10 min, 20 min, 30 min, 1 hr, 3 hr, 6 hr, 9 hr, and 12 hrs post-dose), Day 2 (24 hrs post-dose), Day 3 (48 hrs post-dose)
Population: The PK parameter analysis population included enrolled and treated participants who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
ng/mL | 1.68 (NA) — As only 1 participant was analyzed, geometric coefficient of variation was not calculated. | 84.78 (20) | 183.1 (28) | 496.2 (14) | 814.8 (23)

19. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
ng*hr/mL | 3.82 (NA) — As only 1 participant was analyzed, geometric coefficient of variation was not calculated. | 300.7 (15) | 638.9 (21) | 1557 (19) | 2788 (31)

20. Secondary Outcome: Terminal Elimination Half-Life (t1/2)
Description: t1/2 is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
hour | NA (NA) — Due to low PF-05280602 levels, terminal phase was not well characterized. | 3.533 (0.560) | 3.637 (0.803) | 3.303 (0.638) | 3.580 (0.564)

21. Secondary Outcome: Incremental Recovery (IncRec)
Description: IncRec is the maximum rise in plasma concentration per administered dose.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mcg/kg
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
ng/mL/mcg/kg | 3.48 (NA) — As only 1 participant was analyzed, geometric coefficient of variation was not calculated. | 18.49 (20) | 20.06 (28) | 27.67 (16) | 26.87 (24)

22. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf)
Description: AUCinf is area under the plasma concentration-time curve from time 0 extrapolated to infinite time.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
ng*hr/mL | NA (NA) — Due to low PF-05280602 levels, terminal phase was not well characterized. | 300.7 (15) | 638.9 (21) | 1557 (19) | 2788 (31)

23. Secondary Outcome: Mean Residence Time (MRT)
Description: MRT is AUMCinf/AUCinf, where AUMC is the area under the first moment curve.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
hours | NA (NA) — Due to low PF-05280602 levels, terminal phase was not well characterized. | 7.948 (1.786) | 5.697 (0.727) | 4.963 (0.741) | 5.087 (0.649)

24. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
L/kg | NA (NA) — Due to low PF-05280602 levels, terminal phase was not well characterized. | 0.1168 (35) | 0.08060 (24) | 0.05651 (21) | 0.05494 (32)

25. Secondary Outcome: Clearance (CL)
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood (rate at which a drug is metabolized or eliminated by normal biological processes). Clearance obtained after intravenous infusion dose is influenced by the fraction of the dose absorbed.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr/kg
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
L/hr/kg | NA (NA) — Due to low PF-05280602 levels, terminal phase was not well characterized. | 0.01502 (15) | 0.01423 (21) | 0.01149 (20) | 0.01089 (31)

26. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Median (Full Range); unit: hours
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
hours | 0.167 (NA) [0.167 to 0.167] | 0.167 (15) [0.083 to 0.200] | 0.242 (21) [0.117 to 0.367] | 0.142 (20) [0.083 to 0.333] | 0.150 (31) [0.083 to 0.333]

27. Secondary Outcome: Maximum Mean Decrease From Baseline in Prothrombin Time (PT)
Description: PT measures how long it takes blood to clot. Maximum mean decrease from baseline at any time point was reported.
Time Frame: Baseline through Day 15
Population: The safety population included all enrolled participants who received the study drug.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
seconds | -0.70 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | -3.37 (0.372) | -3.80 (0.629) | -3.85 (0.409) | -4.45 (0.493)

28. Secondary Outcome: Maximum Mean Decrease From Baseline in Activated Partial Thromboplastin Time (aPTT)
Description: aPTT is a blood test that characterizes blood coagulation. Maximum mean decrease from baseline at any time point was reported.
Time Frame: Baseline through Day 15
Population: The safety population included all enrolled participants who received the study drug.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
seconds | -1.30 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | -17.93 (8.944) | -24.47 (12.273) | -43.02 (16.541) | -46.85 (12.281)

29. Secondary Outcome: Maximum Mean Increase From Baseline in Thrombin Anti-Thrombin (TAT) Complexes
Description: TAT complex is a parameter of coagulation and fibrinolysis. The normal reference range of values for TAT is 1 to 4.1 mcg/L. Elevated TAT concentrations may signify predisposition to thrombosis. Maximum mean increase from baseline at any time point was reported.
Time Frame: Baseline through Day 3
Population: The safety population included all enrolled participants who received the study drug. The 'Number of Participants Analyzed' is the number of evaluable participants for this measure.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 5 | 6 | 6
mcg/L | 3.70 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 23.82 (51.130) | 4.72 (5.282) | 5.52 (6.530) | 22.47 (28.010)

30. Secondary Outcome: Maximum Mean Increase From Baseline in Prothrombin Fragments 1+2
Description: Prothrombin fragment 1+2 is a coagulation factor, released when prothrombin is cleaved by activated Factor X. Elevated plasma levels of prothrombin fragment 1+2 indicate high risk of thrombosis. Maximum mean increase from baseline at any time point was reported.
Time Frame: Baseline through Day 3
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: picomoles per liter (pmol/L)
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 5 | 6 | 6
picomoles per liter (pmol/L) | 38.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 31.8 (30.56) | 66.4 (84.73) | 76.7 (28.27) | 238.3 (162.22)

31. Secondary Outcome: Maximum Mean Increase From Baseline in D-Dimers
Description: D-dimer is an indicator of fibrin formation and its subsequent lysis and is a useful biomarker representing overall activation of blood coagulation. Maximum mean increase from baseline at any time point was reported.
Time Frame: Baseline through Day 15
Population: The safety population included all enrolled participants who received the study drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
ng/mL | 240.0 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 75.0 (103.68) | 28.3 (173.60) | 88.3 (123.36) | 238.3 (285.06)

32. Secondary Outcome: Maximum Mean Increase From Baseline in Endogenous Thrombin Potential (ETP)
Description: ETP was evaluated using a Thrombin Generation Assay (TGA), a validated automated ex-vivo assay that measures the ability of plasma to generate thrombin. Thrombin generation curves are generated and calculated using dedicated software. ETP is the area under the thrombin generation curve and represents the total amount of generated thrombin. Maximum mean increase from baseline at any time point was reported.
Time Frame: Baseline through Day 3
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: nanomolar*minute (nM*min)
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 5 | 6 | 6
nanomolar*minute (nM*min) | 13.400 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 212.643 (77.3337) | 186.196 (147.6925) | 287.173 (421.1883) | 522.758 (94.0122)

33. Secondary Outcome: Maximum Mean Decrease From Baseline in Thrombin Generation Lag Time
Description: The lag time is defined as the time to reach one sixth of the peak height and is a measure of the initiation phase. It is equivalent to the clotting time. Maximum mean decrease from baseline at any time point was reported.
Time Frame: Baseline through Day 3
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 5 | 6 | 6
minutes | -0.540 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | -6.235 (5.7141) | -7.088 (7.9294) | -13.400 (14.6902) | -2.425 (0.9507)

34. Secondary Outcome: Maximum Mean Increase From Baseline in Peak Thrombin Generation
Description: The peak height is defined as the maximum thrombin concentration produced. Maximum mean increase from baseline at any time point was reported.
Time Frame: Baseline through Day 3
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Nanomolar (nM)
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Number analyzed (Participants) | 1 | 6 | 5 | 6 | 6
Nanomolar (nM) | -0.620 (NA) — As only 1 participant was analyzed, standard deviation was not calculated. | 17.982 (6.0924) | 16.568 (12.9124) | 23.362 (28.4618) | 49.130 (21.0371)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last study drug administration (Day 60)
Arm/Group | PF-05280602 0.5 mcg/kg | PF-05280602 4.5 mcg/kg | PF-05280602 9.0 mcg/kg | PF-05280602 18.0 mcg/kg | PF-05280602 30.0 mcg/kg
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/1 | 5/6 | 5/6 | 3/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05280602 0.5 mcg/kg (N=1) | PF-05280602 4.5 mcg/kg (N=6) | PF-05280602 9.0 mcg/kg (N=6) | PF-05280602 18.0 mcg/kg (N=6) | PF-05280602 30.0 mcg/kg (N=6)
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The protocol was amended to a starting dose of 4.5 mcg/kg. The positive anti-PF-05280602 antibody was cross-reactive with NovoSeven and native Factor VII and the weak positive immune response at Day 60 may represent a false-positive test result.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Catalyst Biosciences has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.